CLINICAL TRIAL: NCT03073421
Title: A Qualitative Evaluation of the "Positive Pregnancy Program", an Inter-professional Multidisciplinary Program for the Care of HIV-positive Pregnant Women
Brief Title: Positive Pregnancy Program
Acronym: P3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-124
Record Dates: First submitted 2017-02-22; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: HIV Positive Pregnant Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIV positive pregnant women (Other): HIV positive pregnant women who took part in the P3 program will take part in a 2-hour qualitative interview.
  Interventions: Other: Qualitative interview

INTERVENTIONS:
Other: Qualitative interview — This interview will be 2 hours in length and will be conducted with a Peer Research Assistant (PRA). The PRAs will be women living with HIV.

SUMMARY:
The Positive Pregnancy Program is an innovative, unique, interprofessional model of care for HIV-positive pregnant women. This program has been in place at St. Michael's Hospital for five years. This study is important because it will allow for a critical evaluation of the Program, and to identify strengths and weaknesses. This will in turn provide the opportunity to improve delivery of care for HIV positive women.

DETAILED DESCRIPTION:
The aim of the P3 program is to provide supportive and comprehensive care from a variety of perspectives, including medical, social, and psychological. The premises on which the program are built include: a commitment to the respect, confidentiality, dignity and medical care of clients; health promotion; normalizing the care of HIV-positive pregnant women; knowledge translation; and the intentions to build a model of care that is transferable to other clinicians and to other conditions.

During antenatal visits, pregnant women are seen by a multidisciplinary team of professionals including an Obstetrician, Midwife, Prenatal Nurse and Social Worker. Different rooms are used for routine antenatal care maneuvers and for consultation and counseling. The Midwife attends the births of the women in the program, and does home post partum care visits. Care is provided that is patient- and family-centered. Partners are invited to attend as many visits as the couple wishes. Because of this team approach, significantly more time is spent with each woman than would occur at a routine prenatal visit.

The patient population at the St. Michael's clinic is largely made up of immigrant women. Many of these women are refugees, and have fled conflict zones or wars to come to Canada. More than 50% have lived in Canada for less than five years. Many of these women are marginalized, and may not access care elsewhere. They have many issues beyond HIV, and some of the social determinants of health that we observe during their time in the program include issues surrounding housing, finance, immigration, legal issues, social support, co-morbid conditions and substance use.

Since the launch of the program, there has been a rapid increase in the number of women attending each year. The program has also attracted significant attention, both from within the medical and health care communities and beyond.

This study seeks to determine if women cared for in the Positive Pregnancy Program will have a high degree of satisfaction with this model of care.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive pregnant women who took part in P3 program

Exclusion Criteria:

* HIV negative
* did not take part in P3 program

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 25 (Actual)
Dates: Start 2012-06-29 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Degree of satisfaction with P3 program during antenatal period | 36 weeks gestation
  A qualitative 2 hour interview will be conducted with HIV positive pregnant women taking part in the P3 program. The first interview will be timed to occur late in the third trimester, at approximately 36 weeks gestation. This interview will allow an evaluation of women's experiences during antenatal care. The second interview will occur in the post partum period, and will be timed to coincide with the post partum visit at six weeks after birth. This interview will allow an evaluation of women's experiences in the hospital, during labour and delivery, and on the post partum floor.
Post-partum degree of satisfaction with P3 program | 6 weeks post-partum
  The second interview will occur in the post partum period, and will be timed to coincide with the post partum visit at six weeks after birth. This interview will allow an evaluation of women's experiences in the hospital, during labour and delivery, and on the post partum floor.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yudin, MD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No